CLINICAL TRIAL: NCT00542698
Title: Changing Activity Behavior With Glucose Sensor Feedback
Brief Title: Changing Physical Activity Behavior in Individuals With Type 2 Diabetes Using Counceling and Information From Continuous Glucose Monitoring
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Nursing Research (NINR) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00004009; NIH: F31 NR008818-01A1
Record Dates: First submitted 2007-10-10; First posted 2007-10-11 (Estimated); Last update posted 2007-10-11 (Estimated); Status verified 2007-10

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes Mellitus; Glucose Monitor graphs; Physical Activity
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

ARMS (2):
- Control (No Intervention): Control group uses 90 minutes of standard diabetes education/ 7 days using the International Diabetes Center curriculum & update phone call at 4 weeks.
- Intervention (Experimental): Interventional group received standard diabetes education, CGMS monitor, and extra educational topics including CGMS counceling.
  Interventions: Behavioral: Effect of Physical Activity on Type II Diabetes Mellitus

INTERVENTIONS:
Behavioral: Effect of Physical Activity on Type II Diabetes Mellitus — Reviewing participants and a role model's continuous glucose monitor graphs, discussing benefits of physical activity and setting physical activity goals.
  Arms: Intervention

SUMMARY:
The purpose of this study was to develop a nurse counseling intervention to increase physical activity behavior in people with type 2 diabetes and to improve their health

DETAILED DESCRIPTION:
Diabetes affects 20.8 million Americans and is the fifth leading cause of death in the United States. Although physical activity is a cornerstone in the treatment of diabetes, it is difficult to change physical activity behaviors and up to 60% of individuals with diabetes do not participate in regular physical activity. The use of a nurse counseling intervention based on established behavior change theory with technology-derived graphical representations of glucose information created a unique opportunity to test the feasibility of motivating people with type 2 diabetes to change physical activity behaviors. The consent form described the study protocol, participant expectations, benefits, risks, and the process of maintaining participant confidentiality.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Type 2 Diabetes Mellitus
* Three month blood sugar test (HbA1c) > 7.5%
* Not receiving insulin to manage diabetes
* Not engaged in a physical activity program more than 2 days per week
* Able to read and speak English

Exclusion Criteria:

* Not able to walk ¼ mile in 10 minutes
* Taking glucocoricoids
* Serious health problems, such as heart problems, found on examination.

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2004-07; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
increased physical activity | 8 Weeks

SECONDARY OUTCOMES:
BP, BMI, & HgA1c (a long term measure of blood glucose) | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nancy A Allen, Ph.D., Principal Investigator — University of Massachusetts Worcester Medical School
Locations (2):
- United States (2):
  - Berkshire Health System, Pittsfield, Massachusetts
  - Baystate Health System, Springfield, Massachusetts

REFERENCES:
- [Result] Abstract -OR 27: Effect of Counseling with Continuous Glucose Monitoring on Physical Activity Behaviors June 2006, Oral Presentation for American Diabetes Association 66th Scientific Session, Washington D.C